CLINICAL TRIAL: NCT05991440
Title: Racial and Socioeconomic Differences in Chronic Low Back Pain
Brief Title: Examining Racial and Socioeconomic Differences in Chronic Low Back Pain
Acronym: ERASED
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Burel Goodin, Prof of Anesthesiology, Washington University School of Medicine
Other Study IDs: 202306132; R01MD017565 (NIH)
Record Dates: First submitted 2023-07-31; First posted 2023-08-14 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain
Keywords: lower back pain; Race; Socioeconomic
MeSH Terms: conditions — Chronic Pain; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected for analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this research study is to gain a better understanding of how people's racial background and socioeconomic status (e.g., income, education, and employment) impact their experiences of chronic low back pain (cLBP).

ELIGIBILITY:
Inclusion:

* Non-specific cLBP that has persisted for at least 3 months and has resulted in pain on at least half the days in the past 6 months.
* Age 18 - 85; the lower end of this age range was chosen to capture the growing prevalence of young adults with cLBP, and participants over 85 years are increasingly likely to meet one or more exclusion criteria.
* Participants report ethnic group as non-Hispanic and racial group as either Black/African American or White/Caucasian.

Exclusion:

* Low back pain that is attributable to other factors such as ankylosing spondylitis, infection, malignancy, compression fracture of other trauma.
* Systemic rheumatic disease/condition (e.g. rheumatoid arthritis, systemic lupus erythematosus, fibromyalgia).
* Any other chronic pain condition that the participant believes to be more prominent or severe than the low back pain.
* A history of clinically significant surgery to the low back within the past year.
* Uncontrolled hypertension (i.e. SBP/DBP of > 150/95), cardiovascular or peripheral arterial disease.
* Poorly controlled diabetes (HbA1c > 8%).
* Neurological disease (e.g. Parkinson's, multiple sclerosis, epilepsy).
* Serious psychiatric disorder requiring hospitalization within the past 12 months or characterized by active suicidal ideation.
* Diminished cognitive function that would interfere with understanding of study procedures.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study we will incorporate a combination of clinic-based and community-based participant recruitment. Participants will be recruited from the Pain Treatment Clinics at the Wash U Pain Center and VUMC, as well as the surrounding communities in St. Louis and Nashville, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To elucidate racial group disparities in clinical symptoms among NHBs and NHWs with cLBP. | two years
  Clinical pain severity will be observed through quantitative sensory testing and self-reported questionnaires and surveys.
To elucidate racial group disparities in experimental pain sensitivity among NHBs and NHWs with cLBP. | two years
  Quantitative sensory testing equipment and biological markers assayed via blood samples.
To elucidate racial group disparities in psychosocial risk factors, among NHBs and NHWs with cLBP. | two years
  Psychosocial risk factors that will be observed will be greater increases in depressive symptoms, anxiety, and perceived stress, as well as greater social isolation and loneliness through the use of self-reported questionnaires and surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Burel Goodin, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States